CLINICAL TRIAL: NCT02728765
Title: Obstructive Sleep Apnoea and CPAP Treatment Response in Patients With Non-alcoholic Fatty Liver Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof David Shu Cheong Hui, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Fatty liver/OSA/2016
Record Dates: First submitted 2016-03-31; First posted 2016-04-05 (Estimated); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Obstructive Sleep Apnea; Non-alcoholic Fatty Liver Disease
MeSH Terms: conditions — Sleep Apnea, Obstructive; Non-alcoholic Fatty Liver Disease | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- auto CPAP (Active Comparator): Each patient will be interviewed by the physician on duty and invited to participate in the overnight hospital based auto continuous positive airway pressure (CPAP) titration study for 1 night and then commencement of auto CPAP treatment for 6 months.
  Interventions: Device: Continuous positive airway pressure (CPAP)
- Subtherapeutic CPAP (Placebo Comparator): Following detection of obstructive sleep apnea (OSA), each patient randomized to this arm will receive the same CPAP education, mask fitting and short auto CPAP trial for acclimatization but their auto CPAP device will be set at a subtherapeutic level of 4 cmH20 for use at home. The patients randomized to both arms will receive the same general education about OSA, sleep hygiene, avoidance of alcohol, and weight reduction if appropriate.
  Interventions: Device: Continuous positive airway pressure (CPAP)

INTERVENTIONS:
Device: Continuous positive airway pressure (CPAP) — Continuous positive airway pressure (CPAP) is the gold standard treatment for patients with obstructive sleep apnea (OSA). In a previous trials comparing therapeutic CPAP vs subtherapeutic CPAP, CPAP could reduce 24-hour mean blood pressure in mildly sleepy patients with OSA over 3 months whereas our one-year prospective study has shown that reduction of carotid artery intima-media thickness of OSA patients occurred mostly in the first 6 months and was sustained at 12 months in patients with CPAP compliance about 4.7 hours per night.

SUMMARY:
To study the frequency of obstructive sleep apnea (OSA) and continuous positive airway pressure (CPAP) treatment response in patients with non-alcoholic fatty liver disease (NAFLD).

It is hypothesized that CPAP treatment may improve the activities of NAFLD in those with concomitant OSA.

A screening study for OSA followed by a randomized controlled trial of patients with biopsy proven NAFLD being followed up at the hepatology clinic.

Home sleep study, Epworth sleepiness score (ESS), paired proton magnetic resonance spectroscopy (MRS), transient elastography by fibroscan, serum cytokeratin-18 fragment, liver function tests and liver biopsy (only for those with fibroscan evidence of advanced liver fibrosis).

Patients with confirmed symptomatic OSA will be randomized to receive auto CPAP or subtherapeutic CPAP as control over 6 months.

Primary outcome: changes in intrahepatic triglyceride content (IHTG) measured by proton-MRS after 6 months of auto CPAP versus subtherapeutic CPAP.

DETAILED DESCRIPTION:
Investigators propose to screen for obstructive sleep apnea (OSA) by performing a home sleep study on all the patients with biopsy proven non-alcoholic fatty liver disease (NAFLD) being followed up at the Hepatology Clinic, Prince of Wales Hospital, Hong Kong, in phase one of this study. The following conditions have already been excluded as the underlying cause of liver disease in this specific NAFLD cohort: history of excessive alcoholic consumption (more than 30 g/day for men and 20 g/day for women), secondary causes of hepatic steatosis (such as chronic use of systemic corticosteroids), positive hepatitis B surface antigen, anti-hepatitis C virus antibody, or histological evidence of other concomitant chronic liver diseases.

OSA syndrome is defined by apnoea-hypopnoea index (AHI) of 5 per hours or more of sleep plus excessive daytime sleepiness or two of the following symptoms: choking or gasping during sleep, recurrent awakenings from sleep, unrefreshed sleep, daytime fatigue, and impaired concentration. All patients with suspected OSA will undergo initial assessment at the respiratory clinic with the Epworth sleepiness score (ESS) and symptoms evaluation. Patients who have ESS score >9 or at least two OSA symptoms as described above will be invited to join phase two of the study. They will be invited to undergo a home sleep study.

Those with biopsy proven NAFLD who have AHI≥ 5/hr will be randomized into either group A ) auto CPAP with range 4-12 cmH20 or group B) Subtherapeutic CPAP with the auto CPAP fixed at 4 cmH20 by a balanced block design by a third party not involved in the trial.

ELIGIBILITY:
Inclusion Criteria:

* symptoms of obstructive sleep apnea with home sleep study showing apnea hypopnea index of 5/hour or more, subjects with non-alcoholic fatty liver disease (NAFLD) diagnosed by liver biopsy.

Exclusion Criteria:

* (a) unstable cardiovascular diseases (e.g. recent unstable angina, myocardial infarction, stroke or transient ischemic attack within the previous 6 months or severe left ventricular failure), (b) neuromuscular disease affecting or potentially affecting respiratory muscles,(c) moderate to severe respiratory disease (i.e. breathlessness affecting activities of daily living) or documented hypoxemia or awake oxygen saturation <92% or (d) psychiatric disease that limits the ability to give informed consent or complete the study, (e) professional drivers, (f) gross structural ear-nose-throat abnormalities (large nasal polyps, gross nasal turbinate hypertrophy or septal deviation and enlarged "kissing" tonsils of significant size) who need early intervention.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-07-05 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
Changes in intrahepatic triglyceride content (IHTG) | 6 months

SECONDARY OUTCOMES:
Changes in Epworth Sleepiness Score | 6 months
Transient elastography by fibroscan | 6 months
Serum cytokeratin-18 fragment | 6 months
Change in non-alcoholic fatty liver disease(NAFLD) activity score | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: David SC Hui, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No